CLINICAL TRIAL: NCT04062214
Title: Engaging Veterans Seeking Service-Connection Payments in Pain Treatment (TRIAL)
Brief Title: Pragmatic RCT of SBIRT-PM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000022664; 4UH3AT009758-03 (NIH); 1UG3AT009758-01 (NIH)
Record Dates: First submitted 2019-08-13; First posted 2019-08-20 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Substance Use Disorders; Pain
MeSH Terms: conditions — Substance-Related Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Participants receive either usual care or study intervention
Who Masked: Outcomes Assessor
Masking Description: Research Assistants collect data from participant interviews at 12 and 36 weeks follow-up. They will be blind to randomization condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT-PM (Experimental): Screening, Brief Intervention and Referral to Treatment for Pain Management (SBIRT-PM) was developed to promote engagement in multi-modal non-pharmacological pain management among compensation-seeking Veterans with chronic pain. In SBIRT-PM, a clinician meets with the Veteran after the compensation examination to address the presenting MSD complaint. The clinician addresses Veterans' motivation for multi-modal pain care, and explains how pain can be managed using a variety of non-pharmacological pain management services. The clinician spells out how those services can be accessed at VA. Using permissive language about how pain is commonly self-medicated with substances, the clinician transitions to inquiries about use of prescription and non-prescription substances. The clinician then attempts to motivate Veterans to change their behavior if they are misusing substances. Thus, SBIRT-PM addresses the Veteran's presenting pain complaint first and nascent substance use subsequently.
  Interventions: Behavioral: SBIRT-PM
- Usual Care (No Intervention): A Veteran who completes a Compensation examination ordinarily has no further treatment, referral or debriefing as part of the Compensation examination. Veterans will be advised that they should continue to pursue whatever counseling they need outside the study.

INTERVENTIONS:
Behavioral: SBIRT-PM — SBIRT-PM involves an initial telephone-delivered session followed by up to three calls to Veterans in a 12-week period to support Veteran engagement in multi-modal non-pharmacological pain care and to motivate those who misuse substances to change this problematic behavior. SBIRT-PM also includes coordination between the SBIRT-PM clinicians and the PACT nurse case manager after the initial session to support these patient outcomes.
  Arms: SBIRT-PM

SUMMARY:
Veterans seeking compensation for musculoskeletal (MSD) conditions often develop chronic pain and are at high risk for substance misuse. The Investigators propose to test the effectiveness and cost-effectiveness of Screening, Brief Intervention and Referral to Treatment for Pain Management (SBIRT-PM), designed to reduce pain and reduce risky substance use, in part by helping Veterans get comprehensive pain treatment. The study will involve clinicians at a single site contacting Veterans throughout New England by phone to deliver SBIRT-PM counseling in a pragmatic, randomized, clinical trial.

DETAILED DESCRIPTION:
In 2015 alone, 97,223 new Veterans under age 35 began receiving compensation for injuries related to their military service. In total, there are 559,999 post-9/11 Veterans being compensated for back or neck conditions, and a partially overlapping 596,250 for limitation of flexion in joints. Veterans seeking compensation for musculoskeletal conditions often develop chronic pain and are at high risk for substance misuse. Early intervention is needed to arrest worsening pain and risky substance use, particularly among post-9/11 Veterans for whom engagement in non-pharmacological pain treatment has the potential to improve their overall quality of life and spare them the complications of opioid treatments. The service-connection application is an ideal point-of contact for initiating early intervention treatments for these at-risk Veterans. The Investigators propose to test the effectiveness and cost-effectiveness of Screening, Brief Intervention and Referral to Treatment for Pain Management (SBIRT-PM), designed to reduce pain and risky substance use. In brief, the counselor explains that treating both physical and psychological aspects of pain leads to the best outcomes, outlines what VA (and non-VA if preferred) services are available to Veterans, explains that substances are sometimes used for pain relief, and segues into traditional SBIRT. SBIRT-PM's efficacy is supported by a completed clinical trial of 101 Veterans applying for service-connection for MSD, and by studies showing the efficacy of SBIRT for people with risky substance use and of Motivational Interviewing for engagement in non-pharmacological pain care.

During a two-years pilot study, the study team prepared SBIRT-PM for implementation by establishing communication (Relational Coordination is the theoretical framework) between the "hub" where the SBIRT-PM clinician is sited and the "spoke" sites, establishing study related procedures, and piloting the intervention at each of the eight VA medical centers in New England.

In this full clinical trial, investigators will randomize 1100 Veterans applying for compensation related to MSD to either SBIRT-PM or Usual Care (UC) across eight VA medical centers in New England. Outcome assessment by phone will occur at 12 and 36-week follow-ups, and will be corroborated with other sources of information ---the electronic health record. Investigators hypothesize that, compared to Usual Care, SBIRT-PM will be more effective and cost-effective in improving Veterans' pain and substance use. Investigators further hypothesize that a mediator of these improvements will be use of non-pharmacological services, as extracted from VA records from structured data fields and from narrative text in the medical record using an innovative natural language processing algorithm. Screening and referral to treatment at service-connection examinations can transform a widely-used point of entry to VA into a health promoting encounter.

ELIGIBILITY:
Inclusion Criteria:

* Post-9/11 Veteran applying for MSD-related compensation, as ascertained from filed claim,
* Reports a score of ≥4 (threshold for moderately severe pain) on the BPI's Pain Severity subscale (average of four pain intensity items);
* Availability of a landline or cellular telephone for SBIRT-PM.

Exclusion Criteria:

* Reports inability to participate during the study enrollment call
* Received three or more non-pharmacological pain treatment modalities within the last 12 weeks from VA.
* Participating in another PMC3 study as evidenced by a research protocol alert for that study at the time the study invitation letter is mailed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rosen, MD, Principal Investigator — Yale University/ VA Connecticut Healthcare System; Steve Martino, PhD, Principal Investigator — Yale University/ VA Connecticut Healthcare System
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - VA Connecticut Healthcare System (VACHS), West Haven, Connecticut
  - VA Maine Healthcare System, Augusta, Maine
  - Edith Nourse Rogers Memorial VA Hospital (VA Bedford), Bedford, Massachusetts
  - VA Boston Healthcare System, Boston, Massachusetts
  - VA Central Western Massachusetts Healthcare System, Leeds, Massachusetts
  - Manchester VA Medical Center, Manchester, New Hampshire
  - Providence VA Medical Center, Providence, Rhode Island
  - White River Junction VA Hospital, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Week 12
Arm/Group | SBIRT-PM | Usual Care
Started | 558 | 543
Completed | 457 | 432
Not Completed | 101 | 111
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 14 | 13
Not completed — Lost to Follow-up | 55 | 68
Not completed — Intermittent missing | 31 | 29
Period: Week 36
Arm/Group | SBIRT-PM | Usual Care
Started | 488 | 461
Completed | 434 | 409
Not Completed | 54 | 52
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 50 | 46
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBIRT-PM | Usual Care | Total
Number analyzed (Participants) | 558 | 543 | 1101
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (11.1) | 38.9 (10.9) | 39.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 82 | 151
  Male | 489 | 461 | 950
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72 | 83 | 155
  Not Hispanic or Latino | 486 | 460 | 946
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 64 | 72 | 136
  White | 443 | 424 | 867
  Unknown/Other | 51 | 47 | 98
Education [Mean (Standard Deviation); unit: years] | 15 (2.4) | 14.7 (2.2) | 14.9 (2.3)
Married [Count of Participants; unit: Participants] | 303 | 276 | 579
Working for pay [Count of Participants; unit: Participants] — Employment pattern over past 12 months has been full- or -part-time work
  Participants | 446 | 427 | 873
Legal Involvement [Count of Participants; unit: Participants] — Participant endorsed either having (1) served time in jail or (2) has pending charges trial or sentence
  Participants | 65 | 65 | 130
BPI-Intensity [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory (intensity) is a measure for assessing clinical pain. There are four pain severity items rated on a 0-10 scale assessing pain in the past 24 hours. A composite score is the mean of the four severity items on a 0-10 scale with higher scores indicating worse pain.
  units on a scale | 5.4 (1.2) | 5.4 (1.3) | 5.4 (1.3)
BPI-Interference [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory (intensity) is a measure for assessing clinical pain. There are seven pain intensity items rated on a 0-10 scale assessing how pain interfered with seven daily activities (including general activity, walking, work, mood, enjoyment of life, relations with others, sleep) in the past 24 hours. A composite score is the mean of the seven interference items on a 0-10 scale with higher scores indicating worse pain interference.
  units on a scale | 5.1 (2.1) | 5.2 (2.3) | 5.2 (2.2)
PEG [Mean (Standard Deviation); unit: units on a scale] — The "Pain, Enjoyment, General Activity" scale assesses pain intensity and interference in the past week with three questions rated on a 0-10 scale. Questions ask about average pain, pain interference with enjoyment of life, and pain interference with general activity. Mean summary score is calculated using the average of the three items (range 0-10) with a high score indicating more pain intensity/interference.
  units on a scale | 5.7 (1.9) | 5.7 (2.0) | 5.7 (2.0)
Has high-impact chronic pain [Count of Participants; unit: Participants] — High impact chronic pain is a three question assessment that asks about pain in the past three months. Questions ask about how often respondent had pain (never, some days, most days, every day), how often pain limited work activities (never, some days, most days, every day), and if respondent was not working or unable to work due to pain (yes, not).
  Participants | 388 | 372 | 760
Impact of COVID on health care access [Count of Participants; unit: Participants] — Respondents were asked how much the COVID pandemic impacted their ability to access healthcare.
  Participants
    Reduced ability to get health care A LOT | 74 | 86 | 160
    Reduced ability to get health care A LITTLE | 127 | 127 | 254
    NOT AFFECTED ability to get health care | 314 | 284 | 598
    IMPROVED ability to get health care | 26 | 33 | 59
    no response | 17 | 13 | 30
Problematic Substance Use (any) [Count of Participants; unit: Participants] — The ASSIST (Alcohol, Smoking and Substance Involvement Screening Test) v3.0 was used to assess problematic substance use. It consists of 8 questions asking about experience with tobacco products, alcoholic beverages, cannabis, cocaine, amphetamine stimulants, inhalants, sedatives, hallucinogens, opioids, and other substances. For each substance endorsed in Q1, scores from Q2-7 are added together to give a specific substance involvement score.
  A specific substance involvement score above 10 (alcohol) or above 3 (all others) indicates problematic use.
  Participants | 277 | 295 | 572
Problematic Tobacco Use [Count of Participants; unit: Participants] — The ASSIST (Alcohol, Smoking and Substance Involvement Screening Test) v3.0 was used to assess problematic substance use. It consists of 8 questions asking about experience with tobacco products, alcoholic beverages, cannabis, cocaine, amphetamine stimulants, inhalants, sedatives, hallucinogens, opioids, and other substances. For each substance endorsed in Q1, scores from Q2-7 are added together to give a specific substance involvement score.
  A specific substance involvement score above 10 (alcohol) or above 3 (all others) indicates problematic use.
  Participants | 189 | 193 | 382
Problematic Alcohol Use [Count of Participants; unit: Participants] — The ASSIST (Alcohol, Smoking and Substance Involvement Screening Test) v3.0 was used to assess problematic substance use. It consists of 8 questions asking about experience with tobacco products, alcoholic beverages, cannabis, cocaine, amphetamine stimulants, inhalants, sedatives, hallucinogens, opioids, and other substances. For each substance endorsed in Q1, scores from Q2-7 are added together to give a specific substance involvement score.
  A specific substance involvement score above 10 (alcohol) or above 3 (all others) indicates problematic use.
  Participants | 69 | 98 | 167
Problematic Cannabis Use [Count of Participants; unit: Participants] — The ASSIST (Alcohol, Smoking and Substance Involvement Screening Test) v3.0 was used to assess problematic substance use. It consists of 8 questions asking about experience with tobacco products, alcoholic beverages, cannabis, cocaine, amphetamine stimulants, inhalants, sedatives, hallucinogens, opioids, and other substances. For each substance endorsed in Q1, scores from Q2-7 are added together to give a specific substance involvement score.
  A specific substance involvement score above 10 (alcohol) or above 3 (all others) indicates problematic use.
  Participants | 117 | 112 | 229
Problematic Use of substance other than tobacco, alcohol, cannabis)) [Count of Participants; unit: Participants] — The ASSIST (Alcohol, Smoking and Substance Involvement Screening Test) v3.0 was used to assess problematic substance use. It consists of 8 questions asking about experience with tobacco products, alcoholic beverages, cannabis, cocaine, amphetamine stimulants, inhalants, sedatives, hallucinogens, opioids, and other substances. For each substance endorsed in Q1, scores from Q2-7 are added together to give a specific substance involvement score.
  A specific substance involvement score above 10 (alcohol) or above 3 (all others) indicates problematic use.
  Participants | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity Subscale of Brief Pain Inventory
Description: Pain Intensity subscale of the Brief Pain Inventory uses a 0-10 numeric rating scale (0=no pain to 10=pain as bad as you can imagine) to measure four pain severity/intensity items: "worst" pain in the last 24 hours, "least" pain in the last 24 hours, "average" pain, and pain right "now". The pain intensity subscale is scored as a composite of the four pain items (mean intensity score).
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 558 | 543
score on a scale
  week 0 | 5.39 [5.28 to 5.49] | 5.39 [5.28 to 5.50]
  week 12 | 5.02 [4.88 to 5.15] | 4.97 [4.81 to 5.14]
  week 36 | 4.60 [4.45 to 4.76] | 4.86 [4.69 to 5.02]

2. Primary Outcome: Change in Number of Problem Substances Measured by the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
Description: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) was developed to detect and manage substance use and related problems. Substance use will be measured over the last 3 months using Version 3.1.After a screening question focusing on substances ever used, the ASSIST consists of 7 questions about use of and consequences of use of each of 11 classes of substances over the preceding three months (including nicotine, THC and medical THC). Scores are generated for each substance that are mapped to a three-point ordinal score of severity: "no need for treatment", "need for a brief intervention" and "need for an intensive intervention". The number of problem substances are defined as the number of substances above the "no intervention" threshold
  *only participants who had a problem substance reported at baseline were analyzed for this outcome
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: # substances that need treatment
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 277 | 295
# substances that need treatment
  week 0 | 1.47 [1.38 to 1.56] | 1.47 [1.38 to 1.57]
  week 12 | 1.32 [1.20 to 1.44] | 1.19 [1.07 to 1.32]
  week 36 | 1.26 [1.12 to 1.39] | 1.19 [1.06 to 1.31]

3. Primary Outcome: Cost-Effectiveness Ratios (ICERs)
Description: Total costs divided by quality-adjusted life years
Time Frame: 36 weeks
Measure: Number; unit: $/Quality-adjusted life years
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 558 | 543
$/Quality-adjusted life years
  VA perspective | -86925 | -86925
  Societal perspective | 129527 | 129527

4. Primary Outcome: Cost-Effectiveness Acceptability Curves (CEACs)
Description: Probability that SBIRT is cost-effective compared to usual care over a range of monetary values that a decision-maker might consider the maximum acceptable to avoid to improve pain
Time Frame: 36 weeks
Measure: Number; unit: cost-effectiveness probability
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 558 | 543
cost-effectiveness probability
  Threshold of $10k/QALY | .83 | .83
  Threshold of $50k/QALY | .73 | .73
  Threshold of $250k/QALY | .29 | .29

5. Secondary Outcome: Non-pharmacological Pain Service Utilization
Description: Number of modalities of non-opioid pain services used will be assessed using a modified version of the Pain Management Collaboratory's "non-pharmacological and self-care approaches" questionnaire. This questionnaire asks about use of a list of 3 pharmacological and 23 non-pharmacological pain treatment modalities. For each modality, respondents indicate if the treatment was used in the past three months, if the treatment was delivered in an individual or group setting or if done on own (self-care), and the number of sessions/visits attended in the past 3 months. Number of non-pharmacological modalities will be summed.
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: # pain treatment modalities used
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 558 | 543
# pain treatment modalities used
  week 0 | 2.72 [2.56 to 2.87] | 2.49 [2.34 to 2.64]
  week 12 | 3.48 [3.28 to 3.68] | 3.31 [3.11 to 3.51]
  week 36 | 3.33 [3.15 to 3.51] | 3.00 [2.80 to 3.20]

6. Secondary Outcome: Pain Interference Subscale of Brief Pain Inventory
Description: Pain interference subscale of Brief Pain Inventory uses a 0-10 numeric rating scale (0=no interference to 10=interferes completely) to measure seven daily activities: general activity, walking, work, mood, enjoyment of life, relations with others, sleep. The pain interference subscale is scored as the mean of the seven interference items. This mean can be used if more than 50% (4/7 items) have been completed on a given administration.
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 558 | 543
score on a scale
  week 0 | 5.15 [4.97 to 5.32] | 5.16 [4.96 to 5.35]
  week 12 | 4.93 [4.73 to 5.14] | 4.78 [4.55 to 5.02]
  week 36 | 4.35 [4.13 to 4.58] | 4.61 [4.38 to 4.84]

7. Secondary Outcome: Overall Health Measured by EQ-5D-5L
Description: The Eq-5D-5L is a standardized measure of health status designed for clinical and economic appraisals. It includes a health scale which asks respondents to rate their health today on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 558 | 543
score on a scale
  week 0 | 65.13 [63.79 to 66.46] | 65.74 [64.25 to 67.23]
  week 12 | 66.72 [65.20 to 68.24] | 68.82 [67.22 to 70.41]
  week 36 | 68.61 [67.11 to 70.11] | 69.20 [67.58 to 70.83]

8. Secondary Outcome: Individual Substances of Misuse Generated by the ASSIST
Description: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) (Version 3.1) measures substance use risk over the last 3 months. It consists of 7 questions about use of and consequences of use for 11 classes of substances (including nicotine, THC and medical THC).
  Scores for each substance are summed and mapped to a three-point ordinal score of severity. Risk scores for alcohol range from 0-39, where a score of 0-10 indicates "no need for treatment", a score of 11-26 indicates "need for a brief intervention" and a score of 27+ indicates "need for an intensive intervention". Risk scores for tobacco range from 0-31, risk scores for all other substances range from 0-39, where a score of 0-3 indicates "no need for treatment", a score of 4-26 indicates "need for a brief intervention" and a score of 27+ indicates "need for an intensive intervention".
  Individual substances rated above the "no intervention" threshold will be analyzed here.
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT-PM | Usual Care
Number analyzed (Participants) | 277 | 295
score on a scale
  Tobacco, week 0 | 14.05 [13.08 to 15.01] | 13.35 [12.34 to 14.35]
  Tobacco, week 12 | 11.48 [10.23 to 12.73] | 11.97 [10.55 to 13.38]
  Tobacco, week 36 | 11.09 [9.75 to 12.42] | 10.80 [9.46 to 12.14]
  Alcohol, week 0 | 19.32 [17.44 to 21.20] | 17.72 [16.38 to 19.06]
  Alcohol, week 12 | 15.81 [13.44 to 18.17] | 13.04 [11.04 to 15.04]
  Alcohol, week 36 | 12.93 [10.61 to 15.24] | 11.82 [9.99 to 13.66]
  Marijuana, week 0 | 9.14 [8.04 to 10.25] | 8.80 [7.98 to 9.62]
  Marijuana, week 12 | 7.83 [6.63 to 9.03] | 6.69 [5.70 to 7.67]
  Marijuana, week 36 | 7.33 [6.21 to 8.45] | 6.51 [5.51 to 7.50]

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | SBIRT-PM | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/558 | 2/543
Serious Adverse Events (participants affected / at risk) | 100/558 | 92/543
Other Adverse Events (participants affected / at risk) | 109/558 | 89/543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBIRT-PM (N=558) | Usual Care (N=543)
Emergency room visit (Musculoskeletal and connective tissue disorders) | 62 (99) | 77 (117) — Emergency room visit for pain condition
Surgery (Musculoskeletal and connective tissue disorders) | 41 (44) | 24 (27) — Surgery for musculoskeletal disorder
Emergency room visit or Hospital Care (Psychiatric disorders) | 5 (5) | 1 (1) — ER visit or Hospital care for substance use condition
Residential treatment (Psychiatric disorders) | 1 (1) | 1 (1) — Residential treatment for substance use condition
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBIRT-PM (N=558) | Usual Care (N=543)
Report of suicidal ideation (Psychiatric disorders) | 109 (176) | 89 (131)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04062214/Prot_SAP_002.pdf
  • Informed Consent Form (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04062214/ICF_001.pdf